CLINICAL TRIAL: NCT07360600
Title: ACT Together: Implementing a Web-Based Program With Brief Coaching for Parents of Children With Disabilities in Pediatric Outpatient Clinics
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: American Occupational Therapy Foundation (Other)
Responsible Party: Principal Investigator, Areum Han, Associate Professor, University of South Florida
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY009450; AOTFIR24Han (Other Grant/Funding Number: American Occupational Therapy Foundation)
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Parents; Children With Disabilities; Stress; Depression
Keywords: Acceptance and Commitment Therapy; web-based intervention; internet-based intervention; occupational therapist; parents; children with disabilities; depressive symptoms; stress; feasibility; acceptability; usability; implementation; mixed methods; Pilot Study; phone coaching
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acceptance and commitment therapy (ACT) group (Experimental): The ACT group will complete the ACT Together program.
  Interventions: Behavioral: ACT Together

INTERVENTIONS:
Behavioral: ACT Together — ACT Together includes six self-paced, weekly web-based ACT modules and six brief coaching sessions delivered after each module by a trained occupational therapist.

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility, usability, and preliminary benefits of implementing ACT Together for parents of children with disabilities in pediatric outpatient clinics. ACT Together includes six self-paced, web-based modules and brief weekly one-on-one coaching sessions led by a trained occupational therapist. The program is based on acceptance and commitment therapy (ACT), which teaches practical skills to help people handle stress and difficult thoughts or feelings while taking steps toward what matters to them.

The main questions this study aims to answer are:

* Can parents and occupational therapists complete the study activities as planned (e.g., module completion, coaching sessions, and surveys)?
* Is the program usable and acceptable/appropriate/feasible to implement in this setting?
* Do parents show improvements in mental health and coping-related outcomes after participating in the program?
* What are the experiences and perspectives of parents and therapists regarding the program?

Parents as participants will:

* Complete six self-paced web-based modules and brief weekly individual coaching sessions with a trained occupational therapist.
* Complete online questionnaires before starting and after completing the program.
* Take part in one online interview about their experiences and perspectives on the program.

Occupational therapists as participants will:

* Complete therapist training materials and deliver brief individual coaching sessions to parent participants, including completing a post-session checklist.
* Complete brief online questionnaires before starting and after delivering the program.
* Take part in one online interview about their experiences and perspectives on the program.

DETAILED DESCRIPTION:
Parents of children with disabilities often experience elevated psychological distress and may face barriers to accessing timely, evidence-based support. ACT Together is a research-developed program designed to support parents' coping and psychological well-being in a scalable format that can be implemented in pediatric outpatient clinic settings. This study will be a one-group, pretest-posttest mixed-methods pilot to evaluate the feasibility and implementation of ACT Together when delivered as (1) self-paced, web-based acceptance and commitment therapy (ACT) modules and (2) brief coaching provided by occupational therapists working in pediatric outpatient clinics. All study activities will be coordinated by the University of South Florida (USF) and will be completed remotely using secure online platforms; coaching sessions will be delivered by phone.

Occupational therapists will be recruited via a study flyer and will complete an online screening process. Eligible therapists will complete electronic informed consent and baseline questionnaires and will then access therapist-specific training materials in Canvas. Parents of children with disabilities will be recruited through clinic-based flyer dissemination (e.g., posting or placing flyers at reception). Interested parents will contact the study team and will complete online screening. Eligible parents will complete electronic informed consent and baseline questionnaires and will then receive access to the parent Canvas course.

ACT Together will include six self-paced, weekly web-based ACT modules and six brief coaching sessions (approximately 15 minutes each) delivered after each module by a trained occupational therapist. The modules will be hosted on the USF Canvas platform. Two separate Canvas courses will be used: a parent course that includes ACT modules and activities for parents, and a therapist course that includes training materials and structured coaching guidance to support delivery of the brief coaching sessions. Coaching sessions will use structured questions and guidance developed for research purposes and are not intended as standard clinical care. Coaching sessions will be conducted by phone at a mutually agreed time between the parent and the participating occupational therapist. Occupational therapists will complete a brief session checklist in Qualtrics after each coaching session to document that required components were delivered; these checklists will be used to calculate session-level coaching fidelity.

Parents will be encouraged to complete approximately one module per week and to participate in a coaching session after each module over approximately 7-8 weeks. Both parents and occupational therapists will complete questionnaires at pretest and posttest. Parent-reported outcomes will include depressive symptoms, anxiety, perceived stress, psychological quality of life, and ACT-related processes (psychological inflexibility, cognitive fusion, and values-based engagement). Posttest implementation measures will capture perceived usability, acceptability, appropriateness, and feasibility (reported separately by parents and therapists).

Both groups will complete a one-time individual interview at posttest to understand user experiences and implementation perspectives and to inform refinement of the program and study procedures. Post-program interviews will be conducted via the HIPAA-compliant version of Microsoft Teams and will be audio recorded. Interviews are expected to last approximately 40 minutes.

The Canvas course will capture program engagement metrics (e.g., logins, time spent, and module completion) and responses to in-program activities for research purposes. Occupational therapist checklists completed after each coaching session will provide implementation documentation and fidelity indicators. Feasibility indicators will include recruitment yield, enrollment, retention, and adherence (completion of modules and coaching sessions).

All data will be collected electronically using university-approved secure platforms (Qualtrics, the ACT Together program hosted on USF Canvas, and HIPAA-compliant Microsoft Teams). ACT Together will not be publicly available and will be accessible only to enrolled participants using study-specific login credentials. Identifying information will be collected only as needed for study operations (e.g., communication and compensation) and will be stored separately from research data. Study data will be stored in secure, access-controlled USF systems (including USF Box), with access restricted to authorized study personnel. Only de-identified, aggregate results will be used for dissemination.

ELIGIBILITY:
Inclusion Criteria (Parents of children with disabilities):

1. Community-dwelling adults (aged ≥18 years) with primary caregiving responsibility for a child with disabilities (aged <18 years) who is enrolled in a participating clinic;
2. Expected to use services at the participating clinic at least once per week over the next three months;
3. Willing to learn strategies to cope with emotions and thoughts; and
4. Have access to a web-enabled device (e.g., smartphone, tablet, laptop, or desktop) with reliable internet access at home or in a public space (e.g., library).

Exclusion Criteria (Parents of children with disabilities):

1. Cognitive, physical, sensory impairments, or language barriers (non-English speaking) that would impede participation;
2. Suicidal intent or suicide attempt(s) within the past six months;
3. Participation in another parent support research study at the time of recruitment; or
4. More than three hospitalizations of either the parent or child within the past year, or other serious health concerns that would interfere with program engagement.

Inclusion Criteria (Occupational therapists):

1. Have three or more years of clinical experience in a pediatric setting and be willing to participate in training, program implementation, and study evaluations; and
2. Currently work in a clinic that serves at least 15 children who attend the clinic at least once per week, ensuring the ability to recruit up to five parents per clinic.

Exclusion Criteria (Occupational therapists): N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | During the recruitment period (up to approximately 6 months)
  Recruitment rate will be calculated as the number of participants enrolled per week (enrolled = provided electronic informed consent and completed the baseline assessment).
Retention | Baseline through post-intervention (approximately 7-8 weeks)
  Retention will be defined as the proportion of enrolled participants who complete the post-intervention assessment.
Web-based module completion | Baseline through post-intervention (approximately 7-8 weeks)
  Web-based module completion will be defined as the number of web-based modules completed (range 0-6 modules).
Coaching session completion | Baseline through post-intervention (approximately 7-8 weeks)
  Coaching session completion will be defined as the number of coaching sessions completed (range 0-6 sessions).

SECONDARY OUTCOMES:
Usability | Post-intervention (approximately 7-8 weeks)
  Usability will be assessed using the System Usability Scale (SUS; 10 items rated 1 = strongly disagree to 5 = strongly agree; total score 0-100).
Acceptability of the program | Post-intervention (approximately 7-8 weeks)
  Acceptability of the program will be assessed using the Acceptability of Intervention Measure (AIM). AIM includes 4 items rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). Mean scale scores will be calculated and reported separately for parents and therapists.
Appropriateness of the program | Post-intervention (approximately 7-8 weeks)
  Appropriateness will be assessed using the Intervention Appropriateness Measure (IAM). IAM includes 4 items rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). Mean scale scores will be calculated and reported separately for parents and therapists.
Feasibility of the program | Post-intervention (approximately 7-8 weeks).
  Feasibility of the program will be assessed using the Feasibility of Intervention Measure (FIM). FIM includes 4 items rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). Mean scale scores will be calculated and reported separately for parents and therapists.
Change in Patient Health Questionnaire-9 (PHQ-9) scores from baseline to post-intervention | Baseline to post-intervention (approximately 7-8 weeks)
  PHQ-9 is a nine-item self-report questionnaire assessing depressive symptoms over the past two weeks, rated from 0 (not at all) to 3 (nearly every day). Total scores range from 0 to 27, with higher scores indicating greater severity of depressive symptoms.
Change in Generalized Anxiety Disorder -7 (GAD-7) scores from baseline to post-intervention | Baseline to post-intervention (approximately 7-8 weeks)
  GAD-7 is a seven-item self-report questionnaire assessing anxiety symptoms over the past two weeks, rated from 0 (not at all) to 3 (nearly every day). Total scores range from 0 to 21, with higher scores reflecting greater anxiety symptoms.
Change in Perceived Stress Scale-10 (PSS-10) scores from baseline to post-intervention | Baseline to post-intervention (approximately 7-8 weeks)
  PSS-10 is a 10-item questionnaire assessing perceived stress. Items are rated from 0 to 4. Total scores range from 0 to 40, with higher scores indicating greater perceived stress.
Change in World Health Organization Quality of Life-BREF (WHOQOL-BREF) Psychological Health domain scores from baseline to post-intervention | Baseline to post-intervention (approximately 7-8 weeks)
  The WHOQOL-BREF Psychological Health domain includes 6 items rated from 1 to 5. Domain scores will be calculated and reported as transformed scores on a 0-100 scale, with higher scores indicating better psychological quality of life.
Change in Acceptance and Action Questionnaire-II (AAQ-II) scores from baseline to post-intervention | Baseline to post-intervention (approximately 7-8 weeks)
  AAQ-II is a 7-item self-report questionnaire measuring psychological inflexibility. Items are rated from 1 to 7. Total scores range from 7 to 49, with higher scores indicating greater psychological inflexibility.
Change in Cognitive Fusion Questionnaire-7 (CFQ-7) scores from baseline to post-intervention | Baseline to post-intervention (approximately 7-8 weeks)
  CFQ-7 is a 7-item self-report questionnaire measuring cognitive fusion. Items are rated from 1 to 7. Total scores range from 7 to 49, with higher scores indicating a higher degree of cognitive fusion.
Change in Engaged Living Scale-9 (ELS-9) scores from baseline to post-intervention | Baseline to post-intervention (approximately 7-8 weeks)
  ELS-9 is a 9-item self-assessment instrument measuring clarity and engagement with personal values. Items are rated from 1 to 5. Total scores range from 9 to 45, with higher scores indicating increased clarity and engagement with personal values.

OTHER OUTCOMES:
User experiences | Post-intervention (approximately 7-8 weeks)
  Individual interviews (~40 minutes) will be conducted via videoconference to explore experiences among parents (e.g., perceived impact, usability/access, and suggestions for improvement) and therapists (e.g., training, coaching session delivery, and suggestions for improvement).
Coaching session fidelity | Immediately after each coaching session, throughout the intervention period (approximately weeks 1-6) per parent participant
  After each coaching session, occupational therapists complete a module-specific fidelity checklist (item rating: 0 = Not completed, 1 = Partially completed, 2 = Completed). For each session, a fidelity percentage will be calculated as: (sum of item scores ÷ maximum possible score for that module) × 100. Higher percentages indicate greater fidelity to the coaching protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Areum Han, PhD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No